## Effect of High Rebound Mattress Toppers on Sleep and Sleep-Related Symptoms

Statistical Analysis Plan NCT03055156

October 13, 2020

SPSS Statistics for Macintosh, version 26 (IBM corp, Armonk, NY) was used for all analysis. To compare topper effects on sleep [TST, SE, SL, WASO, % of stages of Wake, REM, N1, N2, N3 out of TST], sleep related-factors [Position change frequencies, AHI, and heart rate], and VAS, independent sample t-tests were used.

Topper effects on Core body temperature (CBT) was analyzed using two-way mixed method ANOVA with time and topper type as effects. Topper effects on Mean EEG delta spectral power per second over 90 mins was analyzed using independent sample t tests for each 90 min time bin from lights off (i.e. 0-90min, 90-180 min, 180-270 min, 270-360min).

Significance levels for all analysis were set to p=0.05.